CLINICAL TRIAL: NCT05319509
Title: Pilot Study of Virtual Reality Therapy for Students With Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jack Tsai, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-21-0935
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Anxiety
Keywords: virtual reality; college students
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- gameChange (Experimental)
  Interventions: Device: gameChange

INTERVENTIONS:
Device: gameChange — Staff will explain the rationale behind gameChange, and briefly explain the different scenarios: a doctor's office, a waiting room, a pub, a café, a grocery store, a public street and a bus. Each scenario contains five levels, each increasing with anxiety stimuli and certain tasks the participant must complete. The participant will put on the Oculus headset, and go through a preliminary orientation game. The headset will be casted to an external monitor. Once they start gameChange, it will take the participants to the virtual therapist's room. They will be asked to choose which scenario they would like to participate in first and will complete all five levels for one scenario. Research staff will be taking event sampling-style observations of the participant. After completion of the levels, the participant will return to the virtual therapist's room for debriefing, and then will be asked to exit the game.

SUMMARY:
The purpose of this study is to assess changes in self-reported anxiety over the course of six virtual reality (VR) sessions and to assess changes in academic self-efficacy, as well as examine the feasibility and acceptability of a relatively short and time intensive VR intervention (i.e.,six sessions over the course of three weeks) for reducing anxiety symptoms in college students.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in The University of Texas Health Science Center School of Public Health San Antonio regional campus
* competent in English
* total score of at least 3 on the Generalized Anxiety Disorder (GAD-2)

Exclusion Criteria:

* Currently receiving psychological treatment for anxiety symptoms, or has received treatment in the last year.
* Report photosensitive epilepsy.
* Report stereoscopic vision or balance problems

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in state anxiety as assessed by the Liebowitz Social Anxiety Scale-Self Report version (LSAS-SR) | before first session in week 1, before third session in week 2 and before sixth session in week 3
  The LSAS-SR questionnaire is composed of 24 items divided into 2 subscales, 13 concerning performance anxiety, and 11 pertaining to social situations. The 24 items are first rated on a Likert Scale from 0(none) to 3(severe) on fear felt during the situations, and then the same items are rated from 0(never)-3(usually)regarding avoidance of the situation. Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points. Score of 30 or less indicates social anxiety disorder(SAD) is unlikely, score of 30-60 shows that SAD is probable and score 60-90 indicates that SAD is highly probable.
Change in depressive symptoms as assessed by score on the Patient Health Questionnaire-4 (PHQ-4) | Baseline(before the first session in week 1)
  The PHQ-4 questionnaire consists of 4 questions and each is rated on a 4 point scale from 0(not at all) to 3(every day) for a maximum score of 12,a higher number indicating a worse outcome.
Change in anxiety related behaviors such as rate of speech | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in anxiety related behaviors such as volume of speech | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in anxiety related behaviors such as Negative self-talk | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in anxiety related behaviors such as Utterances about experience | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in anxiety related behaviors such as Laughter | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in Psychomotor agitation such as pacing | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in Psychomotor agitation such as Fidgeting | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in Psychomotor agitation such as Rubbing hands/neck/head | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide
Change in physiology such as perspiration | Week 1(session1 and session 2), week 2( session 3 and session 4), week 3 (session 5 and session 6)
  Anxiety-related behaviors will be recorded using an event sampling observation guide

SECONDARY OUTCOMES:
Change in self-reported academic performance as assessed by the Motivated Strategies for Learning Questionnaire (MSLQ) | before first session in week 1, before third session in week 2 and before sixth session in week 3
  The MSLQ questionnaire consists of 9 questions each one is scored from 1= not at all true of me to 7=very true of me, a higher number indicating a better outcome with a maximum score of 63
change in feasibility as assessed by the rating on a short questionnaire | after the third session in week 2 , after sixth session in week 3
  The usability questionnaire is developed by gameChange about the ease of VR software use, believability of VR environment, and level of engagement. this consists of 5 questions and each one is scored form 1(very difficult) to 5(very easy) for a maximum score of 25, a higher number indicating more easiness in using the VR software
Change in acceptability as assessed by the rating on a short questionnaire | after the third session in week 2 , after sixth session in week 3
  The usability questionnaire is developed by gameChange about the ease of VR software use, believability of VR environment, and level of engagement. this consists of 5 questions and each is scored form 1(strongly disagree) to 5(strongly agree) for a maximum score of 25
Change in perceived presence in the virtual environment (as indicated by continuous score on the Igroup Presence Questionnaire (IPQ) | after the third session in week 2 and the sixth session in week 3
  There are 14 questions and each one is scored form -3 to +3. A total negative score indicates that the participant personally felt very disconnected from VR world, and that they lacked believable presence within world, and rather felt like they were manipulating a machine from an outside perspective.

CONTACTS AND LOCATIONS:
Overall Officials: Tsai Jack, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No